CLINICAL TRIAL: NCT01157884
Title: Change of Body Composition After Kidney Transplantation in Korea
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yon Su Kim, Doctor, Seoul National University Hospital
Other Study IDs: SNUH-001-YH
Record Dates: First submitted 2010-06-09; First posted 2010-07-07 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Kidney Transplantation
Keywords: body composition; obesity; kidney transplantation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — serum: total cholesterol, triglyceride, HDL cholesterol, LDL cholesterol, C-reactive protein (CRP)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney Transplantation

SUMMARY:
The graft survival in kidney transplantation has been improving after the introduction of new immunosuppressive agents. Therefore, other complications after transplantation are concerned; one of those is obesity. Several factors are attributable to obesity in kidney transplant recipients.

The body composition such as fat mass and lean mass is important concept in overweight patients. Some studies have been conducted on the change of body composition in kidney transplants. However, all of them are studied among Caucasians or using dual energy X-ray absorptiometry (DEXA).

In this study, the investigators plan to study the body composition among Asian kidney transplant recipients using the bioelectrical impedance analysis (BIA).

ELIGIBILITY:
Inclusion Criteria:

* aged 20 years and over

Exclusion Criteria:

* history of previous transplantation
* co-transplantation with other organs
* neuropsychological problem with diet (such as anorexia nervosa, bulimia)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: recieved kidney transplantation in the Seoul National University Hospital
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
change of body composition | 2 weeks, 1/3/6/9/12 months after transplantation
  fat mass, lean mass

SECONDARY OUTCOMES:
weight, waist circumference | 2 weeks, 1/3/6/9/12 months after transplantation
cholesterol, CRP | 2 weeks, 1/3/6/9/12 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Yon Su Kim, M.D., Ph.D., Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea